CLINICAL TRIAL: NCT03979482
Title: Skeletal Muscle Mitochondrial Abnormalities and the Metabolic Syndrome in Pulmonary Arterial Hypertension
Brief Title: Skeletal Muscle Mitochondrial Abnormalities and the Metabolic Syndrome in PAH
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Steeve Provencher, Professor, Laval University
Other Study IDs: Syndrome métabolique IRM
Record Dates: First submitted 2019-05-24; First posted 2019-06-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Artery Hypertension
Keywords: skeletal muscle mitochondrial abnormalities; metabolic syndrome; insulin resistance
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAH patients: Male and female subjects, aged between 20 and 60 years old. Absence of obesity/diabètes. PAH patients presenting with metabolic syndrome (MS).
- Sedentary healthy patients: Male and female subjects, aged between 20 and 60 years old. Absence of obesity/diabètes. Healthy but sedentary subjects.

SUMMARY:
Pulmonary arterial hypertension (PAH) is characterized by the progressive increase in pulmonary vascular resistance ultimately leading to right ventricular (RV) failure. Its prevalence is estimated at 40-60 persons per million and predominantly affects people between 20 and 60 years of age. Newly available therapies have improved the 3-year survival to >80%. This improvement in prognosis brings new challenges for clinicians: PAH has changed from a rapidly fatal disease to a chronic disorder with persistent exercise limitation and poor quality of life.

Many observations suggest that exercise limitation in PAH is not simply due to pulmonary hemodynamic impairment, but that other determinants are involved. Interestingly, even in absence of obesity or diabetes, insulin resistance (IR) and metabolic syndrome (MS) are highly prevalent amongst PAH patients and associated with worse outcomes. Indeed, lipid accumulation in skeletal muscle (a feature of IR) is observed in both human and experimental model of PAH, but its impact on skeletal muscle function and thus exercise intolerance in PAH remains elusive.

Over the past years, several pathophysiological pathways activated by MS have been identified, including the downregulation PPARg/PGC1a and the insulin signalling pathways, especially the insulin-receptor substrate 1 (IRS1)-mediated one. The decrease in these axes is associated with lipid accumulation and impaired mitochondrial function. The investigators previously reported in PAH lungs that the downregulation of these pathways contributes to the establishment of the Warburg effect. This metabolic unbalance contributes to pulmonary artery smooth muscle (PASMC) proliferation, and resistance to apoptosis contributing to PA remodelling. The investigators recently documented that PAH skeletal muscles are less perfused and are also characterized by the presence of a Warburg effect. These features were independent of daily life physical activity. Nonetheless, the origin of these abnormalities and their impact on skeletal muscle function have never been studied. The investigators propose to determine whether or not MS seen in PAH patients impairs mitochondrial functions through an IRS1/PPARg/PGC1-dependent mechanism, which will ultimately decrease skeletal muscle function and perfusion, and thus overall exercise capacity.

DETAILED DESCRIPTION:
AIM 1:

To determine whether MS is associated with intramuscular lipid accumulation and impaired skeletal muscle metabolism and perfusion in human PAH.

Rationale: MS and IR are highly prevalent amongst PAH patients even in the absence of obesity and diabetes. There are several lines of evidence in the literature that IR develops with the accumulation of fatty-acid metabolites within insulin-responsive tissues, especially intramyocellular lipid deposition within skeletal muscles. Although the mechanism accounting for lipid accumulation remains elusive, a reduction in lipid oxidation as a result of reduction in mitochondrial density has been proposed. The objectives of Aim 1 are 1) to confirm that PAH patients have increased intramuscular lipid accumulation; 2) to determine whether intramuscular lipid accumulation is associated with impaired skeletal muscle metabolism; 3) to demonstrate that these abnormalities correlate with MS and IR and skeletal muscle function amongst PAH patients.

Experimental approaches: The proposed experiments will be performed on PAH patients (n=10-20) vs. 10 healthy but sedentary subjects matched for age, gender, height and weight (definition based on current recommendations), excluding patients with clinically relevant conditions (e.g. diabetes). These individuals are continuously identified through our systematic plasma biobanking process at the time of right heart catheterization (CER#20735), in which roughly 40% of PAH patients with no obesity/diabetes have MS. In addition to routinely performed analyses: A) blood sample will be drawn for Apolipoprotein A1, Apolipoprotein B, glycated hemoglobin, fasting blood glucose, insulin, adiponectin and leptin. B) MR imaging will be used to assess fat infiltration within the quadriceps muscle, liver and heart (see appendix for details). C) Volitional and non volitional strength and endurance of the dominant quadriceps and VO2peak on cycle ergometer will be assessed, as previously described. D) Percutaneous biopsy specimens of the vastus lateralis muscle of the nondominant leg will be taken. Part of the specimen (≈100mg) will be used for immunohistochemistry fiber typing (ethanol modified technique), capillarisation (quantitative IF using CD31-antibody) and intramyocellular lipid accumulation (Oil red O staining, which stains only the most hydrophobic and neutral lipids, as the investigators previously described. The extracellular flux analyzer Seahorse XF24 will be used on the remaining tissues for real time measurements of oxygen consumption and extracellular acidification rates (glycolysis). To ensure that physical inactivity is not responsible for skeletal muscle lipid accumulation, subjects' daily life physical activities will be objectively quantified during one week using a physical activity monitor (SenseWear® armband).

Interpretation: This multimodality approach will provide comprehensive information to confirm: 1) PAH patients exhibit significant increases in quadriceps muscle lipid accumulation compared to controls; 2) lipid accumulation is increased within the skeletal muscle of PAH patients with MS compared to PAH without MS despite similar levels of physical activity; 3) Lipid accumulation is associated with a reduction in lipid oxidation in vivo; 4) MS/IR and quadriceps muscle function correlate with muscle lipid accumulation/glucose oxidative phosphorylation capacity.

Sample size and analysis: Comparisons between groups will be performed using one-way ANOVA followed by a Tukey-Kramer post-test, after confirmation of normality/equal variances (Levene's test). 10 subjects/group will allow detecting a 1.5±0.5 fold increase in quadriceps muscle lipid accumulation assessed by MRI (primary outcome) with type 1 and 2 errors of 5% and 15%. Based on our preliminary data (Fig.3C), these estimates are conservative.

Alternative approach: Insulin action in the liver has many similarities with insulin action in muscle. Although our proposal focuses on skeletal muscles, ectopic lipid accumulation in the liver is also increasingly recognized as contributing to MS and IR. Since MRI sequences to assess fat infiltration take few minutes only, liver and abdominal adiposity will be assessed during the same exam MR study, as previously described.

AIM 2:

To assess whether IR and MS is related to defects in insulin signalling within PAH skeletal muscles.

Rationale: Numerous studies confirmed a reduction in expression of the peroxisome proliferator-activated receptor (PPAR) γ coactivator 1α in the muscles of patients with type 2 diabetes mellitus, reducing the mitochondrial fatty acid oxidation that promotes the accumulation of diacylglycerol within the muscle. In skeletal muscles, insulin binds to its receptor, activating the receptor tyrosine kinase activity, with subsequent phosphorylation and activation of insulin-receptor substrate 1 (IRS1), ultimately promoting the docking and fusion of glucose transporter (GLUT4)-containing vesicles to the plasma membrane. Accumulation of intracellular diacylglycerol has been shown to specifically activate protein kinases C (PKC) θ, resulting in reduction in tyrosine phosphorylation of IRS1. Consistently, activation of muscle PKCθ and increased serine (inactivation) phosphorylation of IRS1 has been noted in the muscles of individuals with type 2 diabetes mellitus and IR. More recently, the activation of the nuclear respiratory factor-2 (NRF2)-Keap1 pathway (improving mitochondrial oxygen consumption, ATP production and beta-oxidation of fatty acids) has been shown to reduce glucose uptake and IR.

Experimental approaches: The same experimental groups and experimental design as described in aim 1 will be used. A) In order to examine the mechanisms responsible for the reduction of mitochondrial activity in PAH skeletal muscles, the expression of several key transcriptional factors and coregulators that are known to regulate mitochondrial biogenesis will be examined, including PPARγ coactivator 1α (PGC-1α), NRF-2, and mitochondrial transcription factor A (WB and immunoprecipitation assay). Mitochondrial oxidative (citrate synthase, hexokinase) and glycolytic (lactate dehydrogenase, phosphofructokinase) enzymes activity (spectrophotometric techniques) will also be assessed. B) In order to assess the potential role of IRS-1 serine phosphorylation in the pathogenesis of IR, the investigators will also examine IRS-1 serine phosphorylation on several serine residues (Ser307, Ser312, Ser616, Ser636) that have been implicated to interfere with insulin signaling in vitro (WB). PKCθ expression and activity will be assessed using isoform-specific PKC antibodies (WB) and a PKC enzyme assay kit.

Interpretation: The investigators expect to demonstrate that: 1) PAH patients exhibit reduced expression/activation of PPARγ1α, and NRF-2, increased phosphorylation of IRS-1 on critical serine sites and PKCθ activation, leading to a metabolic shift toward glycolysis; 2) these abnormalities dominate amongst PAH-MS patients compared to PAH without MS.

Alternative approach: PKCθ activation has been predominantly associated with MS. However, the same experiments could be done for other members of the PKC gene family. In the event that "classical MS pathways" described above do not account for IR/MS in PAH, the role of skeletal muscle Uncoupling Protein-2 and Sirtuin-3, which have recently been implicated in both IR/MS and PAH, will be explored.

ELIGIBILITY:
Inclusion Criteria:

* PAH patients: Male and female subjects, patients presenting with metabolic syndrome (MS).
* Sedentary healthy patients: Male and female subjects. Healthy but sedentary subjects.

Exclusion Criteria:

* Presence of obesity/diabetes

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The proposed experiments will be performed on PAH patients (n=10-20) vs. 10 healthy but sedentary subjects matched for age, gender, height and weight (definition based on current recommendations), excluding patients with clinically relevant conditions (e.g. diabetes). These individuals are continuously identified through our systematic plasma biobanking process at the time of right heart catheterization (CER#20735), in which roughly 40% of PAH patients with no obesity/diabetes have MS.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Concentration of Intramuscular lipid | Through study completion, an average of 1 year
  MR imaging will be used to assess fat infiltration within the quadriceps muscle, liver and heart.
Level of physical activity | During 1 week
  Subjects' daily life physical activities quantified using a physical activity monitor (SenseWear® armband).
Level of mitochondrial activity in PAH skeletal muscles | Through study completion, an average of 1 year
  The expression of several key transcriptional factors and coregulators that are known to regulate mitochondrial biogenesis will be examined, including PPARγ coactivator 1α (PGC-1α), NRF-2, and mitochondrial transcription factor A (WB and immunoprecipitation assay). Mitochondrial oxidative (citrate synthase, hexokinase) and glycolytic (lactate dehydrogenase, phosphofructokinase) enzymes activity (spectrophotometric techniques) will also be assessed.
Change in serine residues (Ser307, Ser312, Ser616, Ser636) due to IRS-1 serine phosphorylation | Through study completion, an average of 1 year
  Differences in phosphorylation of IRS-1 on critical serine residues (Ser307, Ser312, Ser616, Ser636) that have been implicated to interfere with insulin signaling in vitro will be assessed on skeletal muscle biopsies by Western Blot.
Level of PKCθ activation/activity | Through study completion, an average of 1 year
  Will be assessed on skeletal muscle biopsies using isoform-specific PKC antibodies (WB) and a PKC enzyme assay kit.

CONTACTS AND LOCATIONS:
Overall Officials: Steeve Provencher, MD, MSc, Principal Investigator — IUCPQ - Université Laval
Locations (1):
- IUCPQ-UL, Québec, Quebec, Canada

REFERENCES:
- [Background] Pugh ME, Robbins IM, Rice TW, West J, Newman JH, Hemnes AR. Unrecognized glucose intolerance is common in pulmonary arterial hypertension. J Heart Lung Transplant. 2011 Aug;30(8):904-11. doi: 10.1016/j.healun.2011.02.016. Epub 2011 Apr 13. PMID 21493097
- [Background] Hansmann G, Wagner RA, Schellong S, Perez VA, Urashima T, Wang L, Sheikh AY, Suen RS, Stewart DJ, Rabinovitch M. Pulmonary arterial hypertension is linked to insulin resistance and reversed by peroxisome proliferator-activated receptor-gamma activation. Circulation. 2007 Mar 13;115(10):1275-84. doi: 10.1161/CIRCULATIONAHA.106.663120. Epub 2007 Mar 5. PMID 17339547
- [Background] Malenfant S, Potus F, Fournier F, Breuils-Bonnet S, Pflieger A, Bourassa S, Tremblay E, Nehme B, Droit A, Bonnet S, Provencher S. Skeletal muscle proteomic signature and metabolic impairment in pulmonary hypertension. J Mol Med (Berl). 2015 May;93(5):573-84. doi: 10.1007/s00109-014-1244-0. Epub 2014 Dec 30. PMID 25548805
- [Background] Paulin R, Michelakis ED. The metabolic theory of pulmonary arterial hypertension. Circ Res. 2014 Jun 20;115(1):148-64. doi: 10.1161/CIRCRESAHA.115.301130. PMID 24951764
- [Background] Samuel VT, Petersen KF, Shulman GI. Lipid-induced insulin resistance: unravelling the mechanism. Lancet. 2010 Jun 26;375(9733):2267-77. doi: 10.1016/S0140-6736(10)60408-4. PMID 20609972
- [Background] Morino K, Petersen KF, Dufour S, Befroy D, Frattini J, Shatzkes N, Neschen S, White MF, Bilz S, Sono S, Pypaert M, Shulman GI. Reduced mitochondrial density and increased IRS-1 serine phosphorylation in muscle of insulin-resistant offspring of type 2 diabetic parents. J Clin Invest. 2005 Dec;115(12):3587-93. doi: 10.1172/JCI25151. Epub 2005 Nov 10. PMID 16284649
- [Background] Potus F, Malenfant S, Graydon C, Mainguy V, Tremblay E, Breuils-Bonnet S, Ribeiro F, Porlier A, Maltais F, Bonnet S, Provencher S. Impaired angiogenesis and peripheral muscle microcirculation loss contribute to exercise intolerance in pulmonary arterial hypertension. Am J Respir Crit Care Med. 2014 Aug 1;190(3):318-28. doi: 10.1164/rccm.201402-0383OC. PMID 24977625
- [Background] Mootha VK, Lindgren CM, Eriksson KF, Subramanian A, Sihag S, Lehar J, Puigserver P, Carlsson E, Ridderstrale M, Laurila E, Houstis N, Daly MJ, Patterson N, Mesirov JP, Golub TR, Tamayo P, Spiegelman B, Lander ES, Hirschhorn JN, Altshuler D, Groop LC. PGC-1alpha-responsive genes involved in oxidative phosphorylation are coordinately downregulated in human diabetes. Nat Genet. 2003 Jul;34(3):267-73. doi: 10.1038/ng1180. PMID 12808457
- [Background] Griffin ME, Marcucci MJ, Cline GW, Bell K, Barucci N, Lee D, Goodyear LJ, Kraegen EW, White MF, Shulman GI. Free fatty acid-induced insulin resistance is associated with activation of protein kinase C theta and alterations in the insulin signaling cascade. Diabetes. 1999 Jun;48(6):1270-4. doi: 10.2337/diabetes.48.6.1270. PMID 10342815
- [Background] Yu C, Chen Y, Cline GW, Zhang D, Zong H, Wang Y, Bergeron R, Kim JK, Cushman SW, Cooney GJ, Atcheson B, White MF, Kraegen EW, Shulman GI. Mechanism by which fatty acids inhibit insulin activation of insulin receptor substrate-1 (IRS-1)-associated phosphatidylinositol 3-kinase activity in muscle. J Biol Chem. 2002 Dec 27;277(52):50230-6. doi: 10.1074/jbc.M200958200. Epub 2002 Nov 14. PMID 12006582
- [Background] Holmstrom KM, Baird L, Zhang Y, Hargreaves I, Chalasani A, Land JM, Stanyer L, Yamamoto M, Dinkova-Kostova AT, Abramov AY. Nrf2 impacts cellular bioenergetics by controlling substrate availability for mitochondrial respiration. Biol Open. 2013 Jun 20;2(8):761-70. doi: 10.1242/bio.20134853. eCollection 2013 Aug 15. PMID 23951401
- [Background] Liu Z, Dou W, Ni Z, Wen Q, Zhang R, Qin M, Wang X, Tang H, Cao Y, Wang J, Zhao S. Deletion of Nrf2 leads to hepatic insulin resistance via the activation of NF-kappaB in mice fed a high-fat diet. Mol Med Rep. 2016 Aug;14(2):1323-31. doi: 10.3892/mmr.2016.5393. Epub 2016 Jun 10. PMID 27315552